CLINICAL TRIAL: NCT04558099
Title: Effectiveness of Mindfulness-based Stress Reduction Among Student Teachers
Brief Title: Effectiveness of MBSR Among Student Teachers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 08072020
Record Dates: First submitted 2020-09-16; First posted 2020-09-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2020-07

CONDITIONS: Stress Reduction; Mental Well-being
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBSR (Experimental): MBSR according to international standards (2.5 hours group session once a week in 8 weeks; a silence retreat day; and 45-60 minutes homework six days a week). Content in accordance with MBSR curriculum.
  Interventions: Behavioral: MBSR
- Wait-list control (No Intervention): Usual practice

INTERVENTIONS:
Behavioral: MBSR — Described previously
  Arms: MBSR

SUMMARY:
The aim is to evaluate the effectiveness of Mindfulness-based Stress Reduction among Danish student teachers on their mental well-being. The study is a randomised, controlled trial including 100 teachers.

ELIGIBILITY:
Inclusion Criteria:

* Danish student teacher

Exclusion Criteria:

* acute treatment-demanding clinical depression or a diagnosis of psychosis or schizophrenia
* abuse of alcohol, drugs, medicine

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 67 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-01-12 (Actual); Study Completion 2021-01-12 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale | 2 months from baseline
  Change in perceived stress among the student teachers

SECONDARY OUTCOMES:
Brief Resilience Scale Brief Resilience Scale Brief Resilience Scale Brief Resilience Scale | post MBSR (8 weeks from baseline)
  Change in resilience among the student teachers
Symptom Check List - 5 | post MBSR (8 weeks from baseline)
  Change in symptoms of anxiety and depression among the student teachers
WHO-5 | post MBSR (8 weeks from baseline)
  Change in well-being among the student teachers
Five Facet Mindfulness Questionnaire-15 | post MBSR (8 weeks from baseline)
  Change in mindfulness among the student teachers
Amsterdam Resting State Questionnaire | post MBSR (8 weeks from baseline), 6 and 12 months from baseline
  Change in resting state among the student teachers

CONTACTS AND LOCATIONS:
Overall Officials: Lone Fjorback, PhD, MD, Study Director — Aarhus University, Danish Center for Mindfulness
Locations (1):
- Aarhus University, Department of Clinical Medicine, Danish Center for Mindfulness, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Individual deidentified participant data will be shared by reasonable request, following publication of planned papers.

REFERENCES:
- [Derived] Juul L, Brorsen E, Gotzsche K, Nielsen BL, Fjorback LO. The Effects of a Mindfulness Program on Mental Health in Students at an Undergraduate Program for Teacher Education: A Randomized Controlled Trial in Real-Life. Front Psychol. 2021 Dec 6;12:722771. doi: 10.3389/fpsyg.2021.722771. eCollection 2021. PMID 34938226